CLINICAL TRIAL: NCT02175550
Title: An Open, Prospective, Single Cohort, Multi-centre Study Evaluating the NobelReplace Conical Connection Implants Supported Single -Unit Crowns in the Maxilla.
Brief Title: A 5-year Clinical Evaluation Study on NobelReplace Conical Connection Implants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nobel Biocare (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: T-179
Record Dates: First submitted 2014-06-20; First posted 2014-06-26 (Estimated); Last update posted 2021-03-03 (Actual); Status verified 2021-03

CONDITIONS: Implant; Healthy
Keywords: partially edentulous; maxilla; implants; Conical connection; Nobel Biocare; NobelReplace; Immediate loading; One- stage surgery; Two- stage surgery; supported restoration; patients

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- NR CC (Experimental)
  Interventions: Device: NR CC

INTERVENTIONS:
Device: NR CC

SUMMARY:
A new Nobel Biocare implant, NobelReplace Conical Connection (NR CC) has been developed. The implant is a two piece design to allow both one- and two- stage surgical procedures. The entire implant surface has a porous titanium oxide of approximately 10µm thick (TiUnite) to promote and maintain primary stability, which later on leads to secondary stability.

NR CC implants are used as the foundation for anchoring tooth replacements in either jaw. Restorations range from replacing one single tooth to an entire arch of bridgework. The implants are also intended as retentive elements for overdenture applications.

The present study is designed to evaluate, after the insertion of the NR CC, the marginal bone levels and bone remodelling at the implant sites over various time points up to 5 years. Parameters as soft tissue index, pink aesthetic score (PES) and bleeding on probing (BoP) are as well evaluated together with implant success and survival rate.

Using the OHIP-14 questionnaire patients satisfaction is assessed. The results of this clinical investigation will demonstrate clinical safety and reliability of the NR CC using different treatment options.

ELIGIBILITY:
Inclusion Criteria:

* Obtained informed consent from the subject.
* The subject shall be at least 18 years of age and have passed secession of growth
* The subject must be in such a physical and mental condition that a 5-year follow-up period can be carried out without foreseeable problems. (The patient is committed to the study
* The subject requires single unit implant restoration in the anterior maxilla (FDI 15-25); (ADA 4-13)
* The tooth at the planned study site of interest is extracted or lost at least 2 months before the date of implantation
* Healthy implantation site
* Full mouth bleeding on probing (FMBoP) and full mouth plaque index (FMPI) are both lower or equal to 25%
* The subject shall have a favorable and stable occlusal relationship
* Natural roots are adjacent to the implant site
* Maximum two single unit restorations per patient
* The patient is suitable for a 1-stage surgical procedure
* The patient is suitable for immediate temporization without full occlusal loading
* Subject's acceptance of the scheduled program of clinical and radiographic analysis and maintenance.

Exclusion Criteria:

* Insufficient bone volume at the implant site for placing a NobelReplace CC NP 3.5 implant with a length of at least 8 mm.
* Major bone augmentation procedure at the site of implantation
* Primary stability of the placed implant is ≤35Ncm
* Implant insertion of ≥ 45Ncm
* Acute, untreated periodontitis
* Health conditions, which do not permit the surgical treatment
* Any disorders in the planned implant area such as previous tumors, chronic one disease (such as rheumatoid disease)
* Infections in adjacent tissue of the planned implantation site
* Previous oro-maxillo-facial radiotherapy
* Any ongoing application of interfering medication (steroid therapy, bisphosphonate, etc)
* Alcohol or drug abuse as noted in subject records or in subject history
* Heavy smoking (>10 cigarettes/day)
* Uncontrolled diabetes
* Severe bruxism or other destructive habits
* Pregnant or lactating woman

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 99 (Actual)
Dates: Start 2011-03; Primary Completion 2018-07 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Bone levels and bone remodeling at the implant sites | yearly, from baseline up to 5 years
  The parameter will be measured at 1, 2, 3 and 5 years after implant insertion

SECONDARY OUTCOMES:
Soft Tissue Index | yearly, from baseline up to 5 years
  The parameter will be measured at 1, 2, 3 and 5 years after implant insertion
Pink Aesthetic Score (PES) | yearly, from baseline up to 5 years
  The parameter will be measured at 1, 2, 3 and 5 years after implant insertion
Bleeding on Probing (BoP) | yearly, from baseline up to 5 years
  The parameter will be measured at 1, 2, 3 and 5 years after implant insertion
Patient satisfaction | yearly, from baseline up to 5 years
  Patient satisfaction will be assessed at 1, 2, 3 and 5 years after implant insertion
success and survival rates of implants. | yearly, from baseline up to 5 years
  Success and survival rate will be assessed at 1, 2, 3 and 5 years after implant insertion

REFERENCES:
- [Derived] Fugl A, Zechner W, Pozzi A, Heydecke G, Mirzakhanian C, Behneke N, Behneke A, Baer RA, Nolken R, Gottesman E, Colic S. An open prospective single cohort multicenter study evaluating the novel, tapered, conical connection implants supporting single crowns in the anterior and premolar maxilla: interim 1-year results. Clin Oral Investig. 2017 Jul;21(6):2133-2142. doi: 10.1007/s00784-016-2003-0. Epub 2016 Nov 18. PMID 27864641